CLINICAL TRIAL: NCT05521828
Title: Luteal Phase Ovarian Stimulation With Follitropin Delta and Dydrogesterone: a Randomized Cross Over Pilot Trial
Brief Title: Luteal Phase Ovarian Stimulation With Follitropin Delta and Dydrogesterone
Acronym: LadyDe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CRG UZ Brussel (Other)
Responsible Party: Principal Investigator, Federica Di Guardo, Principal investigator, CRG UZ Brussel
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CS-10459
Record Dates: First submitted 2022-08-25; First posted 2022-08-30 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Oocyte Donors; Oocyte Donation
Keywords: cumulus-oocyte complexes; progestin primed ovarian stimulation; controlled ovarian stimulation; luteal phase ovarian stimulation; follicular phase ovarian stimulation; follitropin delta; dydrogesterone
MeSH Terms: interventions — follitropin delta; Dydrogesterone; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Follitropin delta and dydrogesterone (treatment A followed by treatment B) (Other): Treatment A: Ovarian stimulation is started with daily subcutaneous injections of Follitropin delta (Rekovelle) 12 mcg/daily from day 2 of the follicular phase onwards. Dydrogesterone (Duphaston) 20mg/day will be initiated on stimulation day 7 until the criteria for oocyte trigger are achieved.
  Treatment B: From day 20 of the menstrual cycle onwards, daily subcutaneous injections of Follitropin delta (Rekovelle) 12 mcg/daily will be administered. Dydrogesterone (Duphaston) 20mg/day will be initiated on stimulation day 7 or when serum LH > 10 IU/L until day of trigger.
  For both treatment (A and B) oocyte maturation trigger will be planned when transvaginal ultrasound shows at least 3 follicles >20mm in diameter with a single subcutaneous injection of GnRH agonist (Gonapeptyl 0.2 mg). Oocyte retrieval will be performed 36 hours after trigger. The retrieved cumulus oocyte complexes will be counted, denuded and the number of mature oocytes evaluated.
  Interventions: Drug: Follitropin delta (Rekovelle); Drug: Duphaston; Drug: GnRH agonist (Gonapeptyl)
- Follitropin delta and dydrogesterone (treatment B followed by treatment A) (Other): Treatment B: From day 20 of the menstrual cycle onwards, daily subcutaneous injections of Follitropin delta (Rekovelle) 12 mcg/daily will be administered. Dydrogesterone (Duphaston) 20mg/day will be initiated on stimulation day 7 or when serum LH > 10 IU/L until day of trigger.
  Treatment A: Ovarian stimulation is started with daily subcutaneous injections of Follitropin delta12 mcg/daily (Rekovelle) from day 2 of the follicular phase onwards. Dydrogesterone (Duphaston) 20mg/day will be initiated on stimulation day 7 until the criteria for oocyte trigger are achieved.
  For both treatment (B and A) oocyte maturation trigger will be planned when transvaginal ultrasound shows at least 3 follicles >20mm in diameter with a single subcutaneous injection of GnRH agonist (Gonapeptyl 0.2 mg). Oocyte retrieval will be performed 36 hours after trigger. The retrieved cumulus oocyte complexes will be counted, denuded and the number of mature oocytes evaluated.
  Interventions: Drug: Follitropin delta (Rekovelle); Drug: Duphaston; Drug: GnRH agonist (Gonapeptyl)

INTERVENTIONS:
Drug: Follitropin delta (Rekovelle) — 12 mcg/day will be used for ovarian stimulation in both arms
Drug: Duphaston — 20 mg/day will be used for pituitary suppression in both arms
Drug: GnRH agonist (Gonapeptyl) — (2 ampules:0.2 mg) will be used for ovulation triggering in both arms

SUMMARY:
The last decade has shown a progressive scientific interest for new strategies to improve the outcomes of controlled ovarian stimulation (COS).

Given the fact that interovulatory period has been described to have multiple waves of follicular recruitment, luteal phase ovarian stimulation (LPOS) has been proposed as new protocol for COS, with satisfactory ovarian response and pregnancy outcomes. On the other hand progestin-primed ovarian stimulation (PPOS) is today considered an innovative protocol aiming to achieve multi-follicle recruitment and block the luteinizing hormone (LH) surge through progesterone administration in place of the traditional down regulating or gonadotropin-releasing hormone (GnRH) antagonist. This protocol has been shown to be equally effective as LH suppression with GnRH antagonist reporting equivalent oocyte retrieval rates, endocrine profiles, viable embryo numbers, and pregnancy outcomes. Due to the feasibility and patients-friendly characteristics of PPOS in oocytes donors, the current study aims to investigate the impact on the number of cumulus-oocyte complexes (COCs) when a PPOS protocol is associated to both conventional follicular phase stimulation and LPOS for vitrification of oocytes in oocyte donors. Moreover, it aims to determine whether LPOS using PPOS protocol has comparable outcomes to conventional follicular phase stimulation with PPOS protocol, in oocyte donor patients.

DETAILED DESCRIPTION:
The current study is a single centre randomized, crossover, open label, pilot trial.

The study will be conducted on 50 patients who wish to donate their oocytes. All participants will be informed about the nature of the study and informed consent will be taken from all of them.

Patients will randomly undergo two treatment sequences, treatment sequence 1 and treatment sequence 2. Treatment sequence 1 consists of treatment A followed by treatment B; treat-ment sequence 2 consists of treatment B followed by treatment A. The time-interval between the two treatments (washout period) will be minimum two months after trigger and maximum twelve months. All patients will undergo PPOS: one cycle with follicular phase ovarian stimulation and one cycle with LPOS.

Work up: Complete history, hormonal investigations (FSH, LH, E2, Progesterone, Prolactine, AMH, TSH), Basal transvaginal ultrasound

Treatment A: Ovarian stimulation is started on day 2 of the follicular phase with daily subcutaneous injections of Follitropin delta (Rekovelle) 12 mcg/daily from day 2 of the follicular phase onwards. Dydrogesterone (Duphaston) 20mg/day will be initiated on stimulation day 6 until the day of trigger.

Patients response will be monitored by:

Serum E2, P, FSH, LH and human chorionic gonadotropin (HCG) levels on day 2 of the follicular phase. Patients will be reevaluated on stimulation day 8 every 2 days with ultrasound scan to assess follicular growth and endocrine monitoring with E2, P, FSH and LH levels until the criteria for oocyte trigger are achieved.

Treatment B: From day 20 of the menstrual cycle onwards, daily subcutaneous injections of Follitropin delta (Rekovelle) 12 mcg/daily will be administered.

Dydrogesterone (Duphaston) 20mg/day will be initiated on stimulation day 6 or when serum LH > 10 IU/L until day of trigger.

Patients response will be monitored by:

Serum estradiol E2, P, FSH, LH and HCG levels on day 20 of the follicular phase In case of absence of luteal phase values (progesterone > 1.5 ng/ml) at the blood sample of day 20, stimulation will not be started. In this case, hormonal serum assessment with evaluation of E2, P, FSH and LH levels will be repeated every 2 days until luteal phase values will be achieved, and the stimulation will be started. Patient will be reevaluated on stimulation day 8 every 2 days with ultrasound scan to assess follicular growth and endocrine monitoring with E2, P, FSH and LH levels until the criteria for oocyte trigger are achieved.

Both treatments: Oocyte maturation trigger will be planned when transvaginal ultrasound shows at least 3 follicles >20mm in diameter with a single subcutaneous injection of GnRH agonist (0.2 mg Gonapeptyl). Oocyte retrieval will be performed 36 hours after trigger. The retrieved cumulus oocyte complexes will be counted, denuded and the number of mature oocytes evaluated

Statistical Considerations and Sample size Justification

Fifty - patients (25 for each sequence) need to be included. Considering a dropout rate of about 15%, 66 patients will probably be required to reach an adequate sample size.This is a pilot study, and 50 subjects is considered both practically feasible and sufficient to get reliable results in order to guide further trials in this research area.

The primary endpoint, the total number of cumulus-oocyte complexes, will be compared between the two treatments using an analysis of variance model with subject, period, and treatment as factors. The mean difference between the two treatments and its 95% confidence interval will be estimated from the model.

ELIGIBILITY:
Inclusion Criteria:

* Body mass Index (BMI) ≥18 to < 28
* Signed informed consent
* Regular menstrual cycle length i.e. 24-35 days

Exclusion Criteria:

* Contraindications to the use of gonadotropins
* Endometriosis grade 3-4
* Patients with Anti-mullerian hormone (AMH) <1.1 ng/ml and/or antral follicular count (AFC)<7
* Patients with Follicle Number Per Ovary (FNPO) ≥ 19 and/or AMH >5ng/ml
* Patients under contraception with hormonal intrauterine device (IUD)
* Any untreated endocrine abnormality

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
number of retrieved COCs in both treatment groups | 10-20 minutes after oocyte retrieval
  number of retrieved cumulus-oocyte complexes

SECONDARY OUTCOMES:
Endocrine profile in both treatment groups | through study completion, an average of 1 year
  evaluation of serum E2, FSH, LH, Progesterone
Consumption of gonadotrophins in both treatment groups | through study completion, an average of 1 year
  (mcg) of gonadotrophins used during ovarian stimulation
Duration of ovarian stimulation in both treatment groups | through study completion, an average of 1 year
  days of ovarian stimulation
Days of progestin use in both treatment groups | through study completion, an average of 1 year
  days of progestin use during ovarian stimulation
Total number of MII oocytes in both treatment groups | 1-2 hours after oocyte retrieval
  the number of MII oocytes retrieved that will be assessed after denudation

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Blockeel, Prof, MD, Study Director — Centre for Reproductive Medicine, Universitair Ziekenhuis Brussel, Belgium
Locations (1):
- Brussels Ivf, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baerwald AR, Adams GP, Pierson RA. Ovarian antral folliculogenesis during the human menstrual cycle: a review. Hum Reprod Update. 2012 Jan-Feb;18(1):73-91. doi: 10.1093/humupd/dmr039. Epub 2011 Nov 8. PMID 22068695
- [Background] Baerwald AR, Adams GP, Pierson RA. A new model for ovarian follicular development during the human menstrual cycle. Fertil Steril. 2003 Jul;80(1):116-22. doi: 10.1016/s0015-0282(03)00544-2. PMID 12849812
- [Background] Bosch E, Havelock J, Martin FS, Rasmussen BB, Klein BM, Mannaerts B, Arce JC; ESTHER-2 Study Group. Follitropin delta in repeated ovarian stimulation for IVF: a controlled, assessor-blind Phase 3 safety trial. Reprod Biomed Online. 2019 Feb;38(2):195-205. doi: 10.1016/j.rbmo.2018.10.012. Epub 2018 Dec 14. PMID 30594482
- [Background] Cakmak H, Tran ND, Zamah AM, Cedars MI, Rosen MP. A novel "delayed start" protocol with gonadotropin-releasing hormone antagonist improves outcomes in poor responders. Fertil Steril. 2014 May;101(5):1308-14. doi: 10.1016/j.fertnstert.2014.01.050. Epub 2014 Mar 14. PMID 24636401
- [Background] Chian RC, Chung JT, Downey BR, Tan SL. Maturational and developmental competence of immature oocytes retrieved from bovine ovaries at different phases of folliculogenesis. Reprod Biomed Online. 2002 Mar-Apr;4(2):127-32. doi: 10.1016/s1472-6483(10)61929-3. PMID 12470574
- [Background] Cummins JM, Breen TM, Harrison KL, Shaw JM, Wilson LM, Hennessey JF. A formula for scoring human embryo growth rates in in vitro fertilization: its value in predicting pregnancy and in comparison with visual estimates of embryo quality. J In Vitro Fert Embryo Transf. 1986 Oct;3(5):284-95. doi: 10.1007/BF01133388. PMID 3783014
- [Background] Demirtas E, Elizur SE, Holzer H, Gidoni Y, Son WY, Chian RC, Tan SL. Immature oocyte retrieval in the luteal phase to preserve fertility in cancer patients. Reprod Biomed Online. 2008 Oct;17(4):520-3. doi: 10.1016/s1472-6483(10)60239-8. PMID 18854106
- [Background] Fernandez-Sanchez M, Visnova H, Yuzpe A, Klein BM, Mannaerts B, Arce JC; ESTHER-1 and ESTHER-2 Study Group. Individualization of the starting dose of follitropin delta reduces the overall OHSS risk and/or the need for additional preventive interventions: cumulative data over three stimulation cycles. Reprod Biomed Online. 2019 Apr;38(4):528-537. doi: 10.1016/j.rbmo.2018.12.032. Epub 2018 Dec 23. PMID 30713022
- [Background] Giles J, Alama P, Gamiz P, Vidal C, Badia P, Pellicer A, Bosch E. Medroxyprogesterone acetate is a useful alternative to a gonadotropin-releasing hormone antagonist in oocyte donation: a randomized, controlled trial. Fertil Steril. 2021 Aug;116(2):404-412. doi: 10.1016/j.fertnstert.2021.02.036. Epub 2021 Apr 2. PMID 33814126
- [Background] Guan S, Feng Y, Huang Y, Huang J. Progestin-Primed Ovarian Stimulation Protocol for Patients in Assisted Reproductive Technology: A Meta-Analysis of Randomized Controlled Trials. Front Endocrinol (Lausanne). 2021 Aug 31;12:702558. doi: 10.3389/fendo.2021.702558. eCollection 2021. PMID 34531825
- [Background] Ioannidou PG, Bosdou JK, Lainas GT, Lainas TG, Grimbizis GF, Kolibianakis EM. How frequent is severe ovarian hyperstimulation syndrome after GnRH agonist triggering in high-risk women? A systematic review and meta-analysis. Reprod Biomed Online. 2021 Mar;42(3):635-650. doi: 10.1016/j.rbmo.2020.11.008. Epub 2020 Nov 28. PMID 33483281
- [Background] Kuang Y, Chen Q, Hong Q, Lyu Q, Ai A, Fu Y, Shoham Z. Double stimulations during the follicular and luteal phases of poor responders in IVF/ICSI programmes (Shanghai protocol). Reprod Biomed Online. 2014 Dec;29(6):684-91. doi: 10.1016/j.rbmo.2014.08.009. Epub 2014 Sep 6. PMID 25444501
- [Background] Kuang Y, Hong Q, Chen Q, Lyu Q, Ai A, Fu Y, Shoham Z. Luteal-phase ovarian stimulation is feasible for producing competent oocytes in women undergoing in vitro fertilization/intracytoplasmic sperm injection treatment, with optimal pregnancy outcomes in frozen-thawed embryo transfer cycles. Fertil Steril. 2014 Jan;101(1):105-11. doi: 10.1016/j.fertnstert.2013.09.007. Epub 2013 Oct 23. PMID 24161646
- [Background] Maman E, Meirow D, Brengauz M, Raanani H, Dor J, Hourvitz A. Luteal phase oocyte retrieval and in vitro maturation is an optional procedure for urgent fertility preservation. Fertil Steril. 2011 Jan;95(1):64-7. doi: 10.1016/j.fertnstert.2010.06.064. Epub 2010 Aug 5. PMID 20688325
- [Background] McNatty KP, Hillier SG, van den Boogaard AM, Trimbos-Kemper TC, Reichert LE Jr, van Hall EV. Follicular development during the luteal phase of the human menstrual cycle. J Clin Endocrinol Metab. 1983 May;56(5):1022-31. doi: 10.1210/jcem-56-5-1022. PMID 6403567
- [Background] Nyboe Andersen A, Nelson SM, Fauser BC, Garcia-Velasco JA, Klein BM, Arce JC; ESTHER-1 study group. Individualized versus conventional ovarian stimulation for in vitro fertilization: a multicenter, randomized, controlled, assessor-blinded, phase 3 noninferiority trial. Fertil Steril. 2017 Feb;107(2):387-396.e4. doi: 10.1016/j.fertnstert.2016.10.033. Epub 2016 Nov 29. PMID 27912901
- [Background] Qiao J, Zhang Y, Liang X, Ho T, Huang HY, Kim SH, Goethberg M, Mannaerts B, Arce JC. A randomised controlled trial to clinically validate follitropin delta in its individualised dosing regimen for ovarian stimulation in Asian IVF/ICSI patients. Hum Reprod. 2021 Aug 18;36(9):2452-2462. doi: 10.1093/humrep/deab155. PMID 34179971
- [Background] Yildiz S, Turkgeldi E, Angun B, Eraslan A, Urman B, Ata B. Comparison of a novel flexible progestin primed ovarian stimulation protocol and the flexible gonadotropin-releasing hormone antagonist protocol for assisted reproductive technology. Fertil Steril. 2019 Oct;112(4):677-683. doi: 10.1016/j.fertnstert.2019.06.009. Epub 2019 Jul 29. PMID 31371053
- [Background] Yu S, Long H, Chang HY, Liu Y, Gao H, Zhu J, Quan X, Lyu Q, Kuang Y, Ai A. New application of dydrogesterone as a part of a progestin-primed ovarian stimulation protocol for IVF: a randomized controlled trial including 516 first IVF/ICSI cycles. Hum Reprod. 2018 Feb 1;33(2):229-237. doi: 10.1093/humrep/dex367. PMID 29300975